CLINICAL TRIAL: NCT03945708
Title: Does Whole Blood Adsorber During CPB Reduce the Amount of Vasoactive Drugs Postoperatively in Endocarditis Patients Undergoing Valve Surgery? -a Randomized Controlled Study
Brief Title: Does Whole Blood Adsorber During CPB Reduce Vasoactive Drugs Postoperatively in Endocarditis Patients Undergoing Valve Surgery?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emma Hansson (Other)
Collaborators: CytoSorbents, Inc (Industry)
Responsible Party: Sponsor-Investigator, Emma Hansson, Principal Investigator, Sahlgrenska University Hospital
Organization: Sahlgrenska University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 00001
Record Dates: First submitted 2019-05-09; First posted 2019-05-10 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Infective Endocarditis
MeSH Terms: conditions — Endocarditis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Addition of whole blood adsorber to CPB circuit
  Interventions: Device: CytoSorb
- Control (No Intervention): Standard treatment

INTERVENTIONS:
Device: CytoSorb — Addition of a hemofilter to the cardiopulmonary bypass circuit
  Arms: Treatment

SUMMARY:
The study aims to investigate the effect of addition of an adsorber during cardio pulmonary bypassin patients with infective endocarditis undergoing valve surgery, and if it will decrease the use of vasoactive drugs postoperatively.

ELIGIBILITY:
Inclusion Criteria:

1. Infected endocarditis patients undergoing heart valve surgery.
2. Age over 18 years.

Exclusion Criteria:

1 Declines participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-05-15 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Use of vasoactive substances | 48 hours
  Use of norepinephrine in ICU

SECONDARY OUTCOMES:
Milrinone use | 48 hours
  Amount of milrinone used 24 and 48 hours postoperatively
Chest tube bleeding | 48 hours
  Chest tube output in ml
Blood transfusions | 48 hours
  Transfusion of red blood cells, plasma and platelets

CONTACTS AND LOCATIONS:
Overall Officials: Emma Hansson, MD PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No